CLINICAL TRIAL: NCT06452797
Title: Prognostic Estimates Among ICU Clinicians Caring for Patients Requiring Prolonged Mechanical Ventilation
Brief Title: Prognostic Estimates Among ICU Clinicians
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rush University Medical Center (Other)
Collaborators: University of North Carolina, Chapel Hill (Other)
Responsible Party: Principal Investigator, Jared Greenberg, Principal Investigator, Rush University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 24030801
Record Dates: First submitted 2024-06-05; First posted 2024-06-11 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Mechanical Ventilation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Usual Prognostic Approach (No Intervention): Participants will make form a prognosis using their usual approach
- ProVent-14 Guided Prognostic Approach (Experimental): Participants will be asked to form a prognosis after being provided the patient's ProVent-14 score and its meaning
  Interventions: Behavioral: ProVent-14 score

INTERVENTIONS:
Behavioral: ProVent-14 score — A score to estimate one-year mortality for patients requiring at least 14 days of mechanical ventilation
  Arms: ProVent-14 Guided Prognostic Approach

SUMMARY:
One challenge with decision making for mechanically ventilated is that their prognosis is often uncertain. The ProVent-14 score incorporates clinical variables measured on the 14th day of mechanical ventilation to predict risk of death in one year. The ProVent-14 is easy to calculate has been externally validated. However, it is unclear how often clinicians use the ProVent-14 score to predict long-term outcomes for patients requiring 14 days of mechanical ventilation or if it helps clinicians make more accurate predictions. The purpose of this study is to determine whether ICU clinicians who receive a patient's ProVent-14 score make more accurate predictions for mortality at one year than ICU clinicians who do not.

ELIGIBILITY:
Inclusion Criteria:

* ICU day-shift attending physician, fellow physician, advanced practice provider, or nurse
* Caring directly for a patient who requires invasive mechanical ventilation, 14-16 days after initial intubation, not actively transitioning to comfort-focused care and not with a neuromuscular disease (i.e. ALS) as a cause of respiratory failure.

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 238 (Estimated)
Dates: Start 2024-06-18 (Actual); Primary Completion 2027-06-15 (Estimated); Study Completion 2027-06-15 (Estimated)

PRIMARY OUTCOMES:
Accuracy of one-year mortality rate predictions | One-year after participant enrollment
  Associations between participant predictions (0-100% risk of death) and patient outcomes (death or not) will be determined using logistic regression. Accuracy will be determined by Area Under the Receiver Operating Characteristic (AUROC) analysis.

SECONDARY OUTCOMES:
Confidence in prediction | Upon enrollment
  1-10 scale, 10 being most confident
Comfort communicating prognosis to patient/surrogate | Upon enrollment
  1-10 scale, 10 being most comfortable
Recommendation to transition to comfort-focused care | Upon enrollment
  Yes or No
Accuracy of timing of patient death | One-year after participant enrollment
  Participants who predict the patient has a <50% chance of survival will be asked to predict the month the patient will pass away

OTHER OUTCOMES:
Accuracy of factors influencing prediction | One-year after participant enrollment
  Participants will list up to 5 characteristics of the patient's situation that influenced their prediction

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Rush University Medical Center, Chicago, Illinois
  - Rush Oak Park Hospital, Oak Park, Illinois
  - University of North Carolina, Chapel Hill, North Carolina

IPD SHARING:
Plan to Share IPD: Undecided
to be determined

REFERENCES:
- [Background] Cox CE, White DB, Hough CL, Jones DM, Kahn JM, Olsen MK, Lewis CL, Hanson LC, Carson SS. Effects of a Personalized Web-Based Decision Aid for Surrogate Decision Makers of Patients With Prolonged Mechanical Ventilation: A Randomized Clinical Trial. Ann Intern Med. 2019 Mar 5;170(5):285-297. doi: 10.7326/M18-2335. Epub 2019 Jan 29. PMID 30690645
- [Background] Detsky ME, Harhay MO, Bayard DF, Delman AM, Buehler AE, Kent SA, Ciuffetelli IV, Cooney E, Gabler NB, Ratcliffe SJ, Mikkelsen ME, Halpern SD. Discriminative Accuracy of Physician and Nurse Predictions for Survival and Functional Outcomes 6 Months After an ICU Admission. JAMA. 2017 Jun 6;317(21):2187-2195. doi: 10.1001/jama.2017.4078. PMID 28528347
- [Background] Hough CL, Caldwell ES, Cox CE, Douglas IS, Kahn JM, White DB, Seeley EJ, Bangdiwala SI, Rubenfeld GD, Angus DC, Carson SS; ProVent Investigators and the National Heart Lung and Blood Institute's Acute Respiratory Distress Syndrome Network. Development and Validation of a Mortality Prediction Model for Patients Receiving 14 Days of Mechanical Ventilation. Crit Care Med. 2015 Nov;43(11):2339-45. doi: 10.1097/CCM.0000000000001205. PMID 26247337
- [Background] Buehler AE, Ciuffetelli IV, Delman AM, Kent SA, Bayard DF, Cooney E, Halpern SD, Detsky ME. Contributors to Intensive Care Unit Clinicians' Predictions of Patient Outcomes: A Qualitative Analysis. Am J Crit Care. 2018 Nov;27(6):445-453. doi: 10.4037/ajcc2018100. PMID 30385535